CLINICAL TRIAL: NCT01702311
Title: Benefits of Point-of-Care Glucose Testing and Insulin Supplementation at Bedtime in Insulin Treated Patients With Type 2 Diabetes
Brief Title: Point-of-Care Glucose Testing and Insulin Supplementation
Acronym: POC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Prinicipal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00056041
Record Dates: First submitted 2012-05-08; First posted 2012-10-08 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Diabetes
Keywords: Diabetes; Point of care testing; Hypoglycemia; Basal bolus insulin
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bedtime supplementation (Active Comparator): Patients in this arm will have acqhs (before meals and at bedtime) and 3 am blood glucose testing and will receive sliding scale insulin supplementation as needed.
  Interventions: Drug: Bedtime insulin Aspart (Novolog)
- no bedtime supplementation (No Intervention): Patients in this arm will have ac (before meals), qhs (at bedtime) and 3 am blood glucose testing; however, subjects in this group will NOT receive sliding scale insulin bedtime supplementation.

INTERVENTIONS:
Drug: Bedtime insulin Aspart (Novolog) — Bedtime insulin aspart supplementation based on blood glucose value in the bedtime supplementation arm.
  Other Names: Aspart (Novolog)
  Arms: Bedtime supplementation

SUMMARY:
Capillary point-of-care (POC) testing is advocated as a valuable aid in the management of diabetes and hyperglycemia in the hospital setting. POC testing aims at collecting information on BG levels at different time points during the day in order to assess glycemic control and to guide insulin adjustment/correction doses. Although POC testing provides insights into day-to-day excursions in BG levels, bedtime BG testing triggers the use of insulin supplements that may result in increased frequency of hypoglycemia and is expensive with an estimated annual cost in hospitals of several hundreds of millions of dollars in the U.S. Accordingly, this pilot study aims to assess the utility of POC and insulin supplementation (correction doses) at bedtime in improving glycemic control and in preventing hypoglycemia in non-ICU patients with type 2 diabetes mellitus (T2DM). A total of 250 non-ICU medical and surgical patients treated with basal bolus regimen will undergo POC testing before meals and bedtime (standard of care) and half of the patients will receive insulin correction doses at bedtime for BG > 140 mg/dL following a sliding scale protocol, while the other half will be followed without insulin supplementation at bedtime except for extreme hyperglycemia (BG > 350 mg/dl). Patients will be recruited at Emory University Hospital and Grady Memorial Hospital.

DETAILED DESCRIPTION:
The value of POC testing and use of insulin supplements (correction doses) in particular at bedtime, has not been prospectively evaluated in insulin-treated patients with T2DM. In the non-ICU setting, practice guidelines for the management of hyperglycemia in patients with T2DM favor the use of physiologic (basal-nutritional-correction dose) insulin regimens over sliding scale regular insulin. POC testing is invasive and painful, and has the limitation of providing glycemic profile that is an incomplete picture of BG excursions and is not always an accurate method to monitor glucose compared to laboratory assays in addition to the major expense in health care delivery. The overall objective of this proposal is to conduct the first prospective randomized controlled trial (RCT) to determine the POC glucose testing and use of insulin supplementation at bedtime in improving glycemic control and in preventing hypoglycemia in insulin-treated non-ICU patients with T2DM. The central hypothesis of this proposal is that routine BG measurement and insulin supplementation at bedtime does not improve glycemic control or reduce frequency of hypoglycemia in insulin treated medicine and surgery patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with a known history of T2DM for > 3 months
2. Age 18-80 years
3. Home treatment with either diet alone, any combination of oral antidiabetic agents, non-insulin injectables or insulin therapy
4. BG > 140 mg and < 400 mg/dL without laboratory evidence of diabetic ketoacidosis

Exclusion Criteria:

1. Hyperglycemia without a history of diabetes
2. Acute critical illness admitted to the ICU or expected to require ICU admission
3. Receiving continuous insulin infusion
4. Clinically relevant hepatic disease
5. Patients on corticosteroid therapy
6. Patients with creatinine ≥ 3.5 mg/dl
7. Subjects unable to sign consent
8. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Derived] Vellanki P, Bean R, Oyedokun FA, Pasquel FJ, Smiley D, Farrokhi F, Newton C, Peng L, Umpierrez GE. Randomized controlled trial of insulin supplementation for correction of bedtime hyperglycemia in hospitalized patients with type 2 diabetes. Diabetes Care. 2015 Apr;38(4):568-74. doi: 10.2337/dc14-1796. Epub 2015 Feb 9. PMID 25665812

RESULTS

PARTICIPANT FLOW:
Recruitment Details: General medicine and surgery patients admitted to Emory University and Grady Hospital between May 2012 and December 2013
Groups:
- No Bedtime Supplementation: Patients in this arm will have ac (before meals), qhs (bedtime), and 3 am blood glucose testing; however, subjects in this group will NOT receive sliding scale insulin bedtime supplementation.
Period: Overall Study
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Started | 122 | 113
Completed | 106 | 100
Not Completed | 16 | 13
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Discharge less than 24 hours | 10 | 7
Not completed — Physician Decision | 3 | 4

BASELINE CHARACTERISTICS:
Population: 16 subjects were not included in the data analysis for bedtime supplementation arm 13 subjects were not included in the data analysis for no bedtime supplementation arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation | Total
Number analyzed (Participants) | 106 | 100 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10) | 57 (11) | 57 (11)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 75 | 159
  >=65 years | 22 | 25 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 60 | 54 | 114

OUTCOME MEASURES:

1. Primary Outcome: Mean Fasting Blood Glucose
Description: The primary outcome of the study is to compare differences in mean fasting blood glucose levels between patients receiving insulin supplements at bedtime compared to those without insulin supplementation.
Time Frame: up to 10 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
mg/dL | 162 (44) | 157 (41)

2. Secondary Outcome: Mean Daily BG
Description: Secondary outcomes include differences between treatment groups in any of the following measures: mean daily BG
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | no Bedtime Supplementation | Bedtime Supplementation
Number analyzed (Participants) | 100 | 106
mmol/L | 8.8 (1.7) | 8.7 (1.8)

3. Secondary Outcome: Number of Hypoglycemia (BG < 70 mg/dl)
Description: Secondary outcomes include the number of hypoglycemia (BG < 70 mg/dl) among both the groups.
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Number; unit: number of events
Arm/Group | Bedtime Supplementation | no Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
number of events | 32 | 26

4. Secondary Outcome: Daily Dose of Insulin
Description: Compare the daily dose of insulin used among both groups
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
units/day | 39 (23) | 44 (33)

5. Secondary Outcome: Length of Hospital Stay
Description: Length of hospitalization
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
days | 7 [4 to 13] | 6 [5 to 9]

6. Secondary Outcome: Hospital Mortality
Description: Mortality is defined as death occurring during admission or during the hospital stay
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Number; unit: number of events
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
number of events | 0 | 1

7. Secondary Outcome: Nosocomial Infections (CDC)
Description: Nosocomial infections during hospital stay as per the CDC criteria
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Number; unit: number of events
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
number of events | 0 | 0

8. Secondary Outcome: Pneumonia
Description: Pneumonia (CDC criteria)
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Number; unit: number of events
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
number of events | 1 | 0

9. Secondary Outcome: Bacteremia
Description: Bacteremia with SIRS/Sepsis
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Number; unit: number of events
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
number of events | 0 | 0

10. Secondary Outcome: Participants Will be Followed for the Duration of Hospital Stay, an Expected Average of 6 Days
Description: Respiratory failure, defined as PaO2 value < 60 mm Hg while breathing air or a PaCO2 > 50 mm Hg
Time Frame: daily while in hospital for up to 10 days
Measure: Number; unit: number of events
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
number of events | 1 | 0

11. Secondary Outcome: Acute Renal Failure [Rise >50% of Baseline or Creatinine >2.5 mg/dl]
Description: Acute renal failure [rise >50% of baseline or creatinine >2.5 mg/dl]
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 days
Measure: Number; unit: number of events
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
number of events | 4 | 4

12. Secondary Outcome: Number of BG Within Target
Description: Number of glucose levels within target of 70-140 mg/dl
Time Frame: Participants will be followed over the hospital stay- expected 6 days.
Measure: Number; unit: participants
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Number analyzed (Participants) | 106 | 100
participants | 76 | 74

13. Secondary Outcome: Number of Subjects With BG > 300 mg/dL
Time Frame: Subjects will be followed over the hospital stay: expected 6 days
Measure: Number; unit: participants
Arm/Group | no Bedtime Supplementation | Bedtime Supplementation
Number analyzed (Participants) | 100 | 106
participants | 19 | 13

ADVERSE EVENTS:
Arm/Group | Bedtime Supplementation | No Bedtime Supplementation
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/100
Other Adverse Events (participants affected / at risk) | 32/106 | 26/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bedtime Supplementation (N=106) | No Bedtime Supplementation (N=100)
Hypoglycemic events (Endocrine disorders) | 32 | 26 — blood glucose less than 70 mg/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No